CLINICAL TRIAL: NCT01907087
Title: A Phase 1/2 Open-Label Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Intracerebroventricular BMN 190 in Patients With Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2 (CLN2) Disease
Brief Title: A Phase 1/2 Open-Label Dose-Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Intracerebroventricular BMN 190 in Patients With Late-Infantile Neuronal Ceroid Lipofuscinosis (CLN2) Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190-201
Record Dates: First submitted 2013-07-19; First posted 2013-07-24 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Jansky-Bielschowsky Disease; Batten Disease; Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2; CLN2 Disease
Keywords: Late infantile Neuronal Ceroid Lipofuscinosis Type 2; LINCL; NCL2; CLN2; Jansky-Bielschowsky disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — cerliponase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMN190 (Experimental): recombinant human tripeptidyl peptidase-1 (rhTPP1/cerliponase alfa)
  Interventions: Biological: BMN 190

INTERVENTIONS:
Biological: BMN 190 — 30-300 mg ICV infusion administered every other week for at least 48 weeks.
  Other Names: recombinant human tripeptidyl peptidase-1 (rhTPP1); cerliponase alfa

SUMMARY:
The purpose of this study is to determine whether BMN 190 is safe and effective in the treatment of patients with Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2 (CLN2) disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether BMN 190 is safe and effective in the treatment of patients with Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2 (CLN2) disease. This is an open label Phase 1/2 study conducted in patients with CLN2 disease. Efficacy measures (disease rating scale and MRI) will be compared to a natural history control.

The study will be conducted under cGCP and patients will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of CLN2 determined by TPP1 enzyme activity (dried blood spot) available at study entry. If no genotype information is available, blood will be collected for CLN2 gene analysis at baseline. In addition, blood for TPP1 enzyme activity (dried blood spot) will be collected at baseline to be analyzed centrally
* Has mild to moderate disease documented by a two-domain score of 3- 6 on motor and language domains of the Hamburg Scale, with a score of at least 1 in each of these two domains
* Written informed consent from parent or legal guardian and assent from subject, if appropriate
* Has the ability to comply with protocol requirements, in the opinion of the investigator
* Seizures are stable in the judgement of the investigator

Exclusion Criteria:

* Is less than 3 years old at enrollment
* Is 16 years old or older at enrollement
* Has another inherited neurologic disease, e.g. other forms of CLN or seizures unrelated to CLN2 (patients with febrile seizures may be eligible)
* Has another neurological illness that may have caused cognitive decline (e.g., trauma, meningitis, hemorrhage) before study entry
* Requires ventilation support, except for noninvasive support at night
* Has received stem cell, gene therapy, or ERT for CLN2
* Has contraindications for neurosurgery (e.g., congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Has contraindications for MRI scans (e.g., cardiac pacemaker, metal fragment or chip in the eye, aneurysm clip in the brain)
* Has generalized motor status epilepticus within 4 weeks before the First Dose visit, taking care that status epilepticus is on clinical examination and not only electroencephalogram (EEG) (enrollment may be postponed)
* Has severe infection (e.g., pneumonia, pyelonephritis, or meningitis) within 4 weeks before the First Dose visit (enrollment may be postponed)
* Is prone to complications from intraventricular drug administration, including patients with hydrocephalus or ventricular shunts
* Has known hypersensitivity to any of the components of BMN 190
* Has received any investigational medication within 30 days before the first infusion of study drug or is scheduled to receive any investigational drug other than BMN 190 during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's well being, safety, or clinical interpretability
* Pregnancy any time during the study

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jacoby, Study Director — BioMarin Pharmaceutical
Locations (5):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- University Hamburg-Eppendorf, Hamburg, Germany
- Bambino Gesù Children's Hospital, Rome, Italy
- United Kingdom (2):
  - Guy's & St. Thomas NHS Foundation Trust, London
  - Great Ormond Street Hospital for NHS Foundation Trust, London

REFERENCES:
- [Derived] Specchio N, Gissen P, de Los Reyes E, Olaye A, Camp C, Curteis T, Griffiths A, Butt T, Cohen-Pfeffer J, Slasor P, Sisic Z, Jain M, Schulz A. Exploring concurrent validity of the CLN2 Clinical Rating Scale: Comparison to PedsQL using cerliponase alfa clinical trial data. PLoS One. 2024 May 22;19(5):e0302382. doi: 10.1371/journal.pone.0302382. eCollection 2024. PMID 38776275
- [Derived] Schulz A, Specchio N, de Los Reyes E, Gissen P, Nickel M, Trivisano M, Aylward SC, Chakrapani A, Schwering C, Wibbeler E, Westermann LM, Ballon DJ, Dyke JP, Cherukuri A, Bondade S, Slasor P, Cohen Pfeffer J. Safety and efficacy of cerliponase alfa in children with neuronal ceroid lipofuscinosis type 2 (CLN2 disease): an open-label extension study. Lancet Neurol. 2024 Jan;23(1):60-70. doi: 10.1016/S1474-4422(23)00384-8. PMID 38101904
- [Derived] Gissen P, Specchio N, Olaye A, Jain M, Butt T, Ghosh W, Ruban-Fell B, Griffiths A, Camp C, Sisic Z, Schwering C, Wibbeler E, Trivisano M, Lee L, Nickel M, Mortensen A, Schulz A. Investigating health-related quality of life in rare diseases: a case study in utility value determination for patients with CLN2 disease (neuronal ceroid lipofuscinosis type 2). Orphanet J Rare Dis. 2021 May 12;16(1):217. doi: 10.1186/s13023-021-01829-x. PMID 33980287
- [Derived] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815

RESULTS

PARTICIPANT FLOW:
Groups:
- 300 mg BMN 190: Intracerebroventricular (ICV) infusion every two weeks. This is a study of a single cohort followed for at least 48 weeks at dosing of 300 mg.
  Subjects 1, 2, and 3 were initially assigned to the 30 mg dose, then escalated to 100 mg (and subsequently 300 mg) after data review. Subjects 4, 5, and 6 were initially assigned to the 100 mg dose, then escalated to 300 mg after data review. Subjects 7, 8 and 9 were initially assigned to the 300 mg dose. One patient withdrew after one dose due to unwillingness to comply with study procedures, requiring the addition of a 10th patient to this group. DMC approved full recruitment at the 300 mg dose (n=24) after data review.
Period: Overall Study
Arm/Group | 300 mg BMN 190
Started | 24
Completed | 23
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 300 mg BMN 190: Intracerebroventricular (ICV) infusion every two weeks.
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.3 (1.24)
Age, Customized [Count of Participants; unit: Participants]
  <=5 years | 20
  >5 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Motor-Language (ML) Scale Score During 300 mg Dosing Period
Description: The progression of ceroid lipofuscinosis (CLN2) disease was assessed using adapted motor and language domains of the Hamburg rating scale (ML scale score). Motor and Language are each 0 - 3 point subscales in which 3 represents best function and 0 represents loss of function. The sum of the motor and language scores (ML score, 0-6 points) was used to evaluate the loss of function.
Time Frame: Baseline, Week 49/Last Assessment
Population: Intent to Treat (ITT) Population : all study subjects receiving > 1 dose
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
units on a scale
  Baseline | 3.5 (1.2)
  Last Recorded Observation | 3.1 (1.41)
  Change from Baseline to Last Recorded Observation | -0.4 (0.84)
Statistical Analysis 1: Comparison: 300 mg BMN 190; Responder Analysis using ITT Population: Proportion of Subjects without an Unreversed Two-point Decline or Score of 0 in ML Scale Score at 48 Weeks. A 'response' is defined as the absence of an unreversed two-point decline or score of 0 in the 0-to-6 point CLN2 score at 48 weeks; Test type: Other — Inference is by an exact binomial test of the null hypothesis H0: Prob(response) <= 0.50 vs. the alternative hypothesis H1: Prob(response) > 0.50, where Prob(response) denotes the population probability of a response. The confidence interval is an exact interval with significance level α=0.05; p = 0.0002, exact binomial test; Proportion of responders = 0.87, 95% CI 2-sided [0.66 to 0.97]
Statistical Analysis 2: Comparison: 300 mg BMN 190; Slopes Analysis using ITT Population: Estimated Rate of Decline (300 mg Dosing Period); Test type: Other — Subject rate of decline per 48 weeks is estimated: (baseline CLN2 score - last CLN2 score)/(time elapsed in units of 48 weeks). P-value computed as a two-sided t-test for the hypothesis H0: Rate=2.0 points lost/48 weeks vs. H1: Rate not equal 2.0 points lost/48 weeks; p < 0.0001, t-test, 2 sided; Slope = 0.4, 95% CI 2-sided [0.05 to 0.75], Standard Deviation 0.809

2. Secondary Outcome: Percentage Change From Baseline of Magnetic Resonance Imaging (MRI) at Week 49 During 300 mg Dosing Period: Whole Brain Volume
Description: Percentage changes in whole brain volume from the ITT population for the 300 mg dosing period
Time Frame: Baseline, Week 49
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
percentage change from baseline | -4.4 (8.46)

3. Secondary Outcome: Percentage Change From Baseline of Magnetic Resonance Imaging (MRI) at Week 49 During 300 mg Dosing Period: Volume of Total Grey Matter
Description: Percentage changes in volume of total grey matter from the ITT population for the 300 mg dosing period
Time Frame: Baseline, Week 49
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
percentage change from baseline | -9.7 (8.08)

4. Secondary Outcome: Percentage Change From Baseline of Magnetic Resonance Imaging (MRI) at Week 49 During 300 mg Dosing Period: Total White Matter Volume
Description: Percentage changes in total white matter volume from the ITT population for the 300 mg dosing period
Time Frame: Baseline, Week 49
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
percentage change from baseline | -4.2 (9.58)

5. Secondary Outcome: Percentage Change From Baseline of Magnetic Resonance Imaging (MRI) at Week 49 During 300 mg Dosing Period: Volume of Cerebrospinal Fluid
Description: Percentage changes in volume of cerebrospinal fluid from the ITT population for the 300 mg dosing period
Time Frame: Baseline, Week 49
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
percentage change from baseline | 3.6 (15.3)

6. Secondary Outcome: Percentage Change From Baseline of Magnetic Resonance Imaging (MRI) at Week 49 During 300 mg Dosing Period: Whole Brain Apparent Diffusion Coefficient
Description: Percentage changes in whole brain apparent diffusion coefficient from the ITT population for the 300 mg dosing period
Time Frame: Baseline, Week 49
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | 300 mg BMN 190
Number analyzed (Participants) | 23
percentage change from baseline | 0.02 (0.023)

ADVERSE EVENTS:
Time Frame: Full study period, a mean of 49 weeks
Arm/Group | 300 mg BMN 190
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 16/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg BMN 190 (N=24)
Dental caries (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 6 (8)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Propionibacterium infection (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg BMN 190 (N=24)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Bradycardia (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Constipation (Gastrointestinal disorders) | 7 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 4 (6)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 11 (20)
Developmental delay (General disorders) | 3 (3)
Feeling jittery (General disorders) | 2 (4)
Gait disturbance (General disorders) | 7 (7)
Needle issue (General disorders) | 2 (2)
Pyrexia (General disorders) | 13 (87)
Hypersensitivity (Immune system disorders) | 4 (6)
Conjunctivitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 7 (9)
Oral herpes (Infections and infestations) | 2 (4)
Pharyngitis (Infections and infestations) | 5 (6)
Respiratory tract infection (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 5 (7)
Tonsillitis (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 10 (17)
Urinary tract infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 5 (7)
Fall (Injury, poisoning and procedural complications) | 6 (11)
Head injury (Injury, poisoning and procedural complications) | 2 (3)
Laceration (Injury, poisoning and procedural complications) | 2 (4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
CSF test abnormal (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Atonic seizures (Nervous system disorders) | 2 (4)
Drop attacks (Nervous system disorders) | 2 (2)
Dystonia (Nervous system disorders) | 4 (4)
Epilepsy (Nervous system disorders) | 11 (87)
Extensor plantar response (Nervous system disorders) | 4 (4)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 3 (7)
Hypotonia (Nervous system disorders) | 2 (2)
Language disorder (Nervous system disorders) | 2 (2)
Myoclonus (Nervous system disorders) | 7 (14)
Partial seizures (Nervous system disorders) | 2 (3)
Petit mal epilepsy (Nervous system disorders) | 2 (2)
Pleocytosis (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 14 (110)
Seizure cluster (Nervous system disorders) | 2 (4)
Tremor (Nervous system disorders) | 4 (4)
Abnormal behaviour (Psychiatric disorders) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4)
Irritability (Psychiatric disorders) | 4 (5)
Sleep disorder (Psychiatric disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
10 subjects were assigned in 1 of 3 cohorts in Dose Escalation Period for a 4-22 weeks treatment of 30, 100, and/or 300 mg. 9 subjects completing the Dose Escalation Period, plus 14 new subjects, were administered a stable dose of 300mg for 48 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days